CLINICAL TRIAL: NCT04650061
Title: Study on an Individualized Plan to Improve Patient Compliance to Therapy, Based on Stratification and Use of Telemonitoring for Sleep Apnea With CPAP
Brief Title: PIMA - Individualized Adherence Improvement Plan
Acronym: PIMAGASOXMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Liquide Healthcare Spain (Industry)
Collaborators: Hospital Sao Joao (Other); Hospital Pedro Hispano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 88/CE/JAS
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A multi-centre randomized, controlled trial (RCT)
Who Masked: Participant
Masking Description: The patient is informed that he participates in a study to test the efficacy of different care plans, but he is not informed if he belongs to the experimental or to the control group (standard of care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIMA Group (Experimental): 1. MEntA: Educational & Training Program
  2. Stratification: Identification of Personal Variables (Age, Level of study, Work status, preference of care attention, digital behaviour)
  3. Adherence evaluation: Evaluation of Perceived Competence, Quality of Life, Mood, Activities, Social relations and Social Support
  4. Identification of Care plan and Schedule next visits
  5. Follow-up D21-D90-D120-D180 depending of the care plan, through the channel that belong for each care plan
  Interventions: Behavioral: Motivational Interview (MI) & Adherence Follow-Up
- Control (Active Comparator): 1. Training program
  2. Schedule next visits
  3. Follow-up D21-D90-D120-D180 using the same process: visit at home or phone.
  Interventions: Device: Adherence Follow-Up

INTERVENTIONS:
Behavioral: Motivational Interview (MI) & Adherence Follow-Up — With MI, the key goal is to empower the patient to commit to follow CPAP therapy, while providing empathic support, in a positive atmosphere, and without prejudice. The nurse does not directly advocate for behavior change (i.e. use CPAP as prescribed), but asks key questions to help the patient explore their feelings about the change, weighs the pros and cons of such change, and allows the patient to realize the discrepancy between the current risk (that is, not using CPAP as directed) and the benefits with good adherence.
  Arms: PIMA Group
Device: Adherence Follow-Up — The nurse takes the compliance of the CPAP device, and ask to the patient if he had some problems.
  Arms: Control

SUMMARY:
Continuous positive airway pressure (CPAP) is the first-line treatment for sleep apnoea/hypopnoea syndrome (OSA). The aim of this study is to know the results in adherence to CPAP and health related outcomes in patients with OSA through a comprehensive and multidisciplinary program based on stratification and individualized care plans, including the motivational interview.

Methods: A multicenter randomized controlled trial (RCT) is designed. The control group will follow the usual treatment, while the intervention group (PIMA) will follow the treatment according to the stratification label based on a comprehensive assessment. This label determines a personalized treatment plan for each patient, which includes different channels (home, telephone, care center) and the use of the motivational interview in each of the interventions with the patient. The main outcome was adherence. Secondary outcomes were quality of life, emotional state, activities, social relationships, perceived competence and motivation.

DETAILED DESCRIPTION:
The subjects enrolled in the study are required to have a diagnosis of OSA confirmed by sleep studies with polygraphy (PS) and / or polysomnography(PSG). Prior to enrolment in the study, all patients are informed in detail about the study and signed the consent form to participate. A randomisation process will follow using a random number generator in Statistical Package for the Social Sciences (SPSS) to systematically assign patients to one group or another, with allocation concealment. Responsible for randomization are prescribers.

The control group intervention. The patients will follow the standard of care, which consists of starting therapy in the home, where the nurse perform training in the use of CPAP equipment, mask adjustment, and safety and maintenance instructions. For follow-up, the patient is always visited at home or telephone, with a frequency established by the Portuguese Society of Sleep(Day 7, Day 21 and Day 180). The follow-up procedure consists of reviewing the CPAP hour meter and resolving any incidents that may have arisen, with the necessary corrective actions (change of mask, positive reinforcement, explanation of specific aspects).

The intervention group 'PIMA' (Personalized Adherence Improvement Plan, based on the Spanish acronym), starts the treatment with the educational and training program called MEntA (Motivational Interview for Adherence). MEntA intervention consists of one session lasting approximately 60 minutes, which is divided into two blocks: educational activity and training activity. In the first block, nurse explains the concepts of sleep apnoea and the symptoms, while a patient shows the CPAP treatment and how to optimize this to the fullest. This block is reinforced with documentation in hard copy and digital format. The second block on training activity was based on working with the treatment, equipment, safety, hygiene and advice. MEntA uses the MI to the treatment of OSA with CPAP. In fact, the nurse uses MI not only at the beginning of therapy, but also in every contact that the patient has with the patient throughout the treatment (subsequent follow-up visits, phone calls, etc). For the PIMA group, the nurse was specifically trained to give this intervention to patients, including a training session with a clinical psychologist.

After the educational and training program, the nurse performs the stratification process to know a series of patient characteristics that will allow identifying the best care plan to obtain the best results in adherence and quality of life. The stratification labels that determine the personalized intervention plan are obtained from two types of variables: personal and modulation variables.With the psychological and clinical variables, in this first visit, "predictive" information is obtained on how the patient's adherence will be: high adherence, moderate adherence or low adherence. Taking this information into account, the care plan will start considering how the patient is and their situation with respect to adherence. Low or moderate adherence relative face plans are more intensive than high adherence relative care plans. In follow-up visits (whose frequency depends on the level of adherence), psychological and clinical variables are reviewed and the patient's adherence is added. Depending on their evolution, the care plan is adapted. For patients with low adherence, telemonitoring is used with hours of compliance, the Apnea-hypoanea index(AHI) and air leak.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years, diagnosis of OSA confirmed by sleep studies with polygraphy (PS) and / or polysomnography (PSG)

Exclusion Criteria:

* subjects with obesity-related hypoventilation, severe COPD (chronic obstructive pulmonary disease) , cognitive disorders and those unable to understand the consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-14 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in adherence in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Number of hours using CPAP per night
Change in somnolence in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Residual sleepiness after use of CPAP. Epworth Test
Change in perceived competence in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Self-Efficacy in the CPAP treatment. Perceived Competence Evaluation Questionnaire
Change in Apnea-hypoanea index in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Number of apneas-hypoapneas per night
Change in Air Leaks in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Fly away through the suitcase adaptation of the mask. Measured in liters / per minute

SECONDARY OUTCOMES:
Change in Quality of Life in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Well-Being of the patient related to sleep apnea. Analogical Well-Being in Sleep Apnea Scale
Change in Mood in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Emotional status related to sleep apnea. Ad hoc question
Change in Activities in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Improving general activity after use CPAP. Ad hoc question
Change in Social Relationships in the first 6 months of treatment | Day 21, Day 90, Day 120, Day 180
  Improving general social relations after use CPAP. Ad hoc question

CONTACTS AND LOCATIONS:
Overall Officials: David Rudilla, PhD, Principal Investigator — Air Liquide Healthcare Spain
Locations (1):
- Antonio Ferreira, Avintes, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Publication of results in two phases:
  * National Congress in Portugal
  * Publication in Research Journal
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Q3 - 2021